CLINICAL TRIAL: NCT05439564
Title: Intrathecal Morphine Versus Morphine-dexmedetomidine Combination for Postoperative Pain Control After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Faheem, Assistant professor of anesthesiology, intensive care, and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Intrathecal morphine-precedex
Record Dates: First submitted 2022-06-26; First posted 2022-06-30 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Intrathecal Morphine; Intrathecal Morphine-dexmedetomidine Combination; Postoperative Pain Control; Total Knee Replacement
MeSH Terms: interventions — Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group morphine (Placebo Comparator): Group morphine (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine.
  Interventions: Drug: Morphine
- Group morphine-Dex (Active Comparator): Group morphine-Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine plus 5 mcg of dexmedetomidine.
  Interventions: Drug: Dexmedetomidine; Drug: Morphine
- Group Dex (Active Comparator): Group Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 5 mcg of dexmedetomidine.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Group morphine-Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine plus 5 mcg of dexmedetomidine.
  Other Names: morphine
  Arms: Group morphine-Dex
Drug: Morphine — Group morphine (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine.
  Arms: Group morphine; Group morphine-Dex
Drug: Dexmedetomidine — Group Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 5 mcg of dexmedetomidine.
  Arms: Group Dex

SUMMARY:
Total knee replacement is one of the most painful orthopedic surgical procedures. Patients who undergo total knee replacement are usually older and have limited cardiac and pulmonary reserves. The increased sensitivity of elderly patients to drugs makes it necessary to choose postoperative analgesia agents and methods that have minimal side effects.

Intrathecal injection of morphine to provide postoperative analgesia during the initial 24-h after the operation is a widely used technique, however, opioid therapy is limited because of the side effects (hypotension, pruritus, nausea, urinary retention, respiratory depression) and intolerance.

Alpha-2 adrenergic agonists (clonidine and dexmedetomidine) have pharmacologic characteristics (sedation, hypnosis, anxiolysis, sympatholytic, and analgesia) that make them suitable as adjuvants to multimodal analgesia.

Their anti-nociceptive effect is attributed to the stimulation of a2- adrenoceptors located in the central nervous system.

The rationale for combining analgesics that produce similar therapeutic effects or synergistic interactions is to accentuate the analgesic efficacy and decrease the side effects by permitting dose reduction of each agent. Human studies on the antinociceptive effects of co-administrated intrathecal morphine (ITM) and dexmedetomidine in postoperative pain are still few.

On the other hand, Abdel-Ghaffar et al., results do not support improved analgesia with the combination of intrathecal morphine and dexmedetomidine, despite the absence of significant adverse effects.

We hypothesized that the addition of dexmedetomidine to ITM would improve the quality of perioperative pain control and decrease the side effects of postoperative systemic opioid use.

DETAILED DESCRIPTION:
105 patients, aged >50 years, with ASA Physical Status Class II and III, scheduled for TKR under spinal anesthesia will be included in this study.

105 Patients will be randomly allocated into three equal groups (35 patients each):

* Group morphine (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine.
* Group morphine-Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 0.1 mg of morphine plus 5 mcg of dexmedetomidine.

Group Dex (35 patients): patients will be received given 0.5% heavy bupivacaine (3.5 ml) plus 5 mcg of dexmedetomidine

Measurements:

1. Demographic data as age, BMI, ASA status, duration of surgery
2. During surgery, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate (HR) will be recorded at the 1st, 5th, 15th, 30th, and 60th minutes.
3. Postoperative pain severity assessed by the visual analog score for pain at rest (ranging from 0 to 10, where 0 no pain and 10 maximum pain) will be evaluated postoperatively at 30 min and 2, 4, 6, 12, and 24 h postoperative. Accordingly, the patient is requested to verbally express his degree of pain using this scale. Patients with the visual analog score≥ 4 will be received 3 mg morphine IV and will be recorded. Patients who complained of pain (the visual analog score< 3) and needed analgesics will be treated intravenous infusion every six to eight hours with Diclofenac Na(75mg).
4. The total dose of morphine used postoperatively will be observed and recorded for the 1st, 2nd, 6th, 12th, and 24th postoperative hours.
5. The period from the moment the intrathecal injection will be made postoperatively until the first analgesic became necessary will be recorded
6. Any recorded postoperative complication as sedation, nausea and vomiting, respiratory depression.
7. The patient's level of sedation will be assessed at the same time points using Ramsay Sedation Scale (score 3-4 mean adequate sedation). (17)

ELIGIBILITY:
Inclusion Criteria:

* 105 patients, aged >50 years, with ASA Physical Status Class II and III, scheduled for TKR under spinal anesthesia

Exclusion Criteria:

1. Patients who had bleeding disorders
2. Patients who had heart, liver, or renal failure
3. Patients who had systemic infections or infections of their injection sites
4. Patients with a known allergy to study
5. Patients who had 2nd or 3rd-degree heart block
6. Those with low back pain or other back problems
7. History of drug or alcohol abuse
8. Body mass index (BMI) > 30 kg\m2
9. Patients with psychiatric illnesses that would interfere with perception and assessment of pain.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The onset of pain | upto 24 hours postoperative
  The onset of pain is defined as VAS ≥ 4 within 24 hours

SECONDARY OUTCOMES:
Postoperative pain severity | upto 24 hours postoperative
  VAS ≥ 4 within 24 hours
The amount of additional analgesic required | upto 24 hours postoperative
  Patients with VAS ≥ 4 will be received 3 mg morphine IV. Patients who complained of pain (VAS < 3) and needed analgesics will be treated with intravenous infusion every six to eight hours with Diclofenac Na(75mg).
Postoperative complications | upto 24 hours postoperative
  the incidence of PONV, respiratory depression, and itching.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tantan University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No